CLINICAL TRIAL: NCT00934687
Title: Clostridium Botulinum Type A Neurotoxin Complex for Adjuvant Treatment of Depressive Disorders - a Randomized Controlled Pilot Study
Brief Title: Botulinum Toxin for the Treatment of Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009DR2125; EKBB14/09
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Depression
Keywords: depression; depressive; botulinum; botox
MeSH Terms: conditions — Depression | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clostridium botulinum toxin type A neurotoxin complex (Experimental): A total of 20-50 U of clostridium botulinum toxin type A neurotoxin complex (Allergan) will be injected at four to six sites in the glabella region according to standard protocols of cosmetic botulinum toxin applications.
  Interventions: Drug: clostridium botulinum toxin type A neurotoxin complex
- 0.9% sodium chloride NaCl solution (Placebo Comparator): 0.9% NaCl solution will be injected like the experimental compound
  Interventions: Other: 0.9% NaCl solution

INTERVENTIONS:
Drug: clostridium botulinum toxin type A neurotoxin complex — A total of 20-50 U of clostridium botulinum toxin type A neurotoxin complex (Allergan) will be injected at four to six sites in the glabella region according to standard protocols of cosmetic botulinum toxin applications.
  Other Names: Vistabel; Botox Cosmetic; Botox
  Arms: clostridium botulinum toxin type A neurotoxin complex
Other: 0.9% NaCl solution — 0.9% NaCl solution will be injected in analogy to clostridium botulinum toxin type A neurotoxin complex as a placebo comparator.
  Other Names: NaCl 0.9% B. Braun
  Arms: 0.9% sodium chloride NaCl solution

SUMMARY:
Depression is frequently accompanied by a specific sad facial expression. This expression is in part mediated by the same muscle activity that produces frown lines. Based on the assumption that there is a positive feedback between depressed mood and the correspondent facial muscle activity (facial feedback) the investigators will conduct a randomized controlled pilot study in which the investigators will apply a classical cosmetic treatment of frown lines with injections of botulinum toxin to depressed patients who did not sufficiently respond to antidepressant medication. The investigators hypothesize that this treatment will contribute to the amelioration of depressive symptoms in these patients. This hypothesis is supported by a previous open case series in which remission of depression was reported after such treatment (Finzi and Wasserman, 2006).

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate depression (Ham-D >=15)
* Therapy with one antidepressant for at least four weeks
* at least moderate frown line

Exclusion Criteria:

* Bipolar depression
* Psychiatric comorbidity
* Severe somatic comorbidity
* Pregnancy
* Peculiarities at the injection site
* Psychiatric medication other than one antidepressant
* Specific psychotherapy
* Previous application of botulinum toxin
* Medication interfering with botulinum toxin

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Response rate (reduction in Ham-D score by >30% compared to baseline) | six weeks

SECONDARY OUTCOMES:
Remission rate (number of patients with HAM-D score < 8) | six weeks
Time to response (20% reduction of HAM-D score compared to baseline) | two, four, or six weeks
response by self rating (BDI) | six weeks
need for additional treatment | eight weeks, twelve weeks, or sixteen weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Wollmer, MD, Principal Investigator — Asklepios Klinik Nord - Ochsenzoll, Hamburg/D; Tillmann HC Krüger, MD, Principal Investigator — Medical School HannoverPsychiatry, Social Psychiatry and Psychotherapy, Hannover, Germany
Locations (2):
- Medical School Hannover, Psychiatry, Social Psychiatry and Psychotherapy, Hanover, Germany
- Psychiatry Hospital of the University of Basel, Basel, Switzerland, Basel, Basel Town, Switzerland